CLINICAL TRIAL: NCT04636281
Title: Comparison of Active and Passive Static Stretching in Delayed Onset of Muscle Soreness of Recreational Body Builders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/00719 Riaz Ahmed
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Sports Physical Therapy
Keywords: Active Stretching; PassiveStretching; Recreational body players
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive static stretching exercise (Experimental): Group 1 will receive passive static stretching. All subjects will be assessed before the intervention through likert muscle soreness scale, Numeric Rating Pain Scale and range of motion for Shoulder, elbow, and wrist by a Goniometer. After that all subjects will perform eccentric exhaust weight exercises in the gym of all mentioned joints, three sets at each joint. Before giving the intervention they will assess of all mentioned parameters.
  Interventions: Other: Active and passive static stretching exercises
- Active static stretching (Experimental): Group 2 will receive active static stretching. All subjects will be assessed before the intervention through likert muscle soreness scale, Numeric Rating Pain Scale and range of motion for Shoulder, elbow, and wrist by a Goniometer. After that all subjects will perform eccentric exhaust weight exercises in the gym of all mentioned joints, three sets at each joint. Before giving the intervention they will assess of all mentioned parameters.
  Interventions: Other: Active and passive static stretching exercises

INTERVENTIONS:
Other: Active and passive static stretching exercises — Different group of muscles will be stretched one by one, tricep brachii, bicep brachii, wrist exentsor etc

SUMMARY:
To find out the better treatment options from active and passive static stretching in delayed onset of muscle soreness in recreational body players.

DETAILED DESCRIPTION:
After registering participant's randomization will be done through sealed envelope method and will be allocated in both groups equally. Group 1 will receive passive static stretching while group 2 will receive active static stretching. All subjects will be assessed before the intervention through likert muscle soreness scale, Numeric Rating Pain Scale and range of motion for Shoulder, elbow, and wrist by a Goniometer. After that all subjects will perform eccentric exhaust weight exercises in the gym of all mentioned joints, three sets at each joint. Before giving the intervention they will assess of all mentioned parameters. Group 1 groups will perform passive static stretching and group 2 will perform active static stretching. At the end of the intervention participants will be assessed again using the same parameters. Statistical analysis will be carried out to compare the outcomes measures of both groups.

ELIGIBILITY:
Inclusion Criteria:

* Recreational Body Builders are Included

Exclusion Criteria:

* Individuals with disc herniation and
* Acute muscle soreness are excluded

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 144 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | 8 weeks
  Assesses the subjective intensity of pain; ages 18 and above
Goniometer | 8 weeks
  A goniometer is an instrument which measures the available range of motion at a joint.
  Range of measurements flexion extension, abduction adduction, internal and external rotation, elbow flexion and extension wrist flexion and extension and radial and ulner deviation
Likert muscle Soreness Scale | 8 weeks
  Scale Description 0 An absence of soreness
  1. A light pain felt only when touched / a vague ache
  2. A moderate pain felt only when touched / a slight persistent pain
  3. A light pain when walking up or down stairs
  4. A light pain when walking on a flat surface / painful
  5. A moderate pain, stiffness or weakness when walking / very painful
  6. A severe pain that limits my ability to move

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Karim, PP-DPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Shahif international Gym, Islamabad, Federal
  - Liaqat Gym, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith M. Effect of Myofascial Decompression on Delayed Onset Muscle Soreness Following Exercise-Induced Muscle Damage. 2018.
- [Background] Paulsen G, Mikkelsen UR, Raastad T, Peake JM. Leucocytes, cytokines and satellite cells: what role do they play in muscle damage and regeneration following eccentric exercise? Exerc Immunol Rev. 2012;18:42-97. PMID 22876722
- [Background] Nikolaidis M. The Effects of Eccentric Exercise on Muscle Damage and Blood Redox Status in Men and Women. Journal of Functional Morphology and Kinesiology. 2017;2(2):20.
- [Background] Pearcey GE, Bradbury-Squires DJ, Kawamoto JE, Drinkwater EJ, Behm DG, Button DC. Foam rolling for delayed-onset muscle soreness and recovery of dynamic performance measures. J Athl Train. 2015 Jan;50(1):5-13. doi: 10.4085/1062-6050-50.1.01. Epub 2014 Nov 21. PMID 25415413
- [Background] Jamtvedt G, Herbert RD, Flottorp S, Odgaard-Jensen J, Havelsrud K, Barratt A, Mathieu E, Burls A, Oxman AD. A pragmatic randomised trial of stretching before and after physical activity to prevent injury and soreness. Br J Sports Med. 2010 Nov;44(14):1002-9. doi: 10.1136/bjsm.2009.062232. Epub 2009 Jun 11. PMID 19525241
- [Background] Xie Y, Feng B, Chen K, Andersen LL, Page P, Wang Y. The Efficacy of Dynamic Contract-Relax Stretching on Delayed-Onset Muscle Soreness Among Healthy Individuals: A Randomized Clinical Trial. Clin J Sport Med. 2018 Jan;28(1):28-36. doi: 10.1097/JSM.0000000000000442. PMID 28742609
- [Background] Kanda K, Sugama K, Hayashida H, Sakuma J, Kawakami Y, Miura S, Yoshioka H, Mori Y, Suzuki K. Eccentric exercise-induced delayed-onset muscle soreness and changes in markers of muscle damage and inflammation. Exerc Immunol Rev. 2013;19:72-85. PMID 23977721